CLINICAL TRIAL: NCT04368650
Title: Evaluation of Rhbmp-2 And Sticky Bone in Intrabony Defects - A Randomized Controlled Trial
Brief Title: RhBMP-2 in Intrabony Defects - A Randomized Controlled Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SVS Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, Dr R Viswa Chandra, Primary Investigator, SVS Institute of Dental Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SVSIDS/PERIO/4/2017
Record Dates: First submitted 2020-04-23; First posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Periodontitis
Keywords: Sticky bone; Intrabony defects; Regeneration
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: Randomization involved the computerized generation of the allocation sequence in random permuted blocks (block randomization) and blinding was ensured by assigning the block of sites to study groups according to the specified sequence by a second operator who coded the two treatment sites selected from every patient by the first operator into the following groups
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Main treatment group (Experimental): The in situ BMP-2 gel was prepared to a concentration of approximately 0.5 μg/ml and were stored at 4oC. The gel was then dispensed at site of interest in the study.
  Interventions: Drug: BMP-2
- Control (Active Comparator): In patients selected for control group, after degranulation, sticky bone was used to fill the defect. The surgical site was protected and covered using a periodontal dressing.
  Interventions: Procedure: PRF

INTERVENTIONS:
Drug: BMP-2 — lyophilized Human Bone Morphogenetic Protein-2 was used as an active drug.
  Other Names: Experimental group
  Arms: Main treatment group
Procedure: PRF — For the preparation of sticky bone, the patient's venous blood is collected and centrifuged at 2400rpm for 2min which leads to two different layers in the vacutainer the upper autologous fibrin glue (AFG) and the lower RBC portion, the upper AFG is mixed with a particulate bone graft (hydroxyapatite). Within 5-10 min fibrin meshwork was formed
  Other Names: Sticky bone group
  Arms: Control

SUMMARY:
This study evaluated the regenerative potential of rhBMP-2 gel in intrabony defects when compared to sticky bone (control).

DETAILED DESCRIPTION:
It was done in 40 subjects who were evaluated for a period of 6 months. the results were evaluated clinically (CAL, PPD) and radiographically (bone fill) and after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy male and female patients age 20-55 years with intrabony defects and probing pocket depth of ≥5mm after initial therapy were included in the study.

Exclusion Criteria:

* Medically compromised patients, Subjects who underwent radiotherapy or chemotherapy and smokers were excluded.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
bone fill | 6 months
  bone fill evaluation done after 6 months by using ImageJ® software

CONTACTS AND LOCATIONS:
Locations (1):
- SVS Institute of Dental Sciences, Mahabubnagar, Hyderabad, Andhra Pradesh, India

IPD SHARING:
Plan to Share IPD: No
No plans to share IPD.